CLINICAL TRIAL: NCT03164096
Title: The Effect of Body Mass Index, Intra-abdominal Pressure, Abdominal Girth and Waist Circumference on Sensory Block Level After Single-shot Spinal Anesthesia for Cesarean Section
Brief Title: The Effect of Some Parturients' Characteristics on Sensory Block Level After Spinal Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: obstanesth
Record Dates: First submitted 2017-05-20; First posted 2017-05-23 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia, Obstetrical
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: evaluating relationship of sensory level and other patient factors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intrathecal bupivacaine (Experimental): intrathecal bupivacaine hydrochloride 0.5%,12.5mg
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — intrathecal bupivacaine will be used for spinal anesthesia in obstetric patients undergoing C-section
  Other Names: intrathecal bupivacaine

SUMMARY:
Although the exact mechanism remains unknown, the association of pregnancy and decreased local anesthetic requirement is clear. demonstrated that more local anesthetic is required for cesarean section under combined spinal-epidural anesthesia in preterm compared with term patients.

DETAILED DESCRIPTION:
However, in pregnant patients, venous engorgement is prominent in the supine but not the lateral position, which suggests direct compression of the inferior vena cava by the gravid uterus. Second, an increase in intraabdominal pressure may affect the retroperitoneal area and may cause inward movement of soft tissue in the intervertebral foramina. Recent magnetic resonance imaging studies in pregnant patients, although without intraabdominal pressure measurements, suggested the latter because they showed limited contact of engorged veins along the dural sac which may therefore not be responsible for compression of the dura.

If elevated intraabdominal pressure contributes to high anesthetic spread during pregnancy, one would expect a relationship between intraabdominal pressure and maximum sensory block level.

ELIGIBILITY:
Inclusion Criteria:

* adult female partner
* aged 18 to 40 years.
* scheduled for elective cesarean section.

Exclusion Criteria:

* Patients with coagulopathy or under anti-coagulation therapy.
* Gastrointestinal disease,
* motion sickness.
* diabetes mellitus.
* Patients with preeclampsia,

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
sensory level | from allocation until 24 hours post-operative
  effect of different parameters in sensory level
motor block | from allocation until 24 hours post-operative
  effect of different parameters in motor level

SECONDARY OUTCOMES:
hypotension | from allocation until 24 hours post-operative
  incidence of hypotension after spinal anesthesia
vasopressor consumption | from allocation until 24 hours post-operative
  total dose of ephedrine consumed by the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided